CLINICAL TRIAL: NCT03686228
Title: Treatment of No-option CLI Patients by G-CSF-mobilized Autologous Peripheral Blood Mononuclear Cells
Brief Title: Treatment of No-option CLI by G-CSF-mobilized PB-MNC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SI016033012/2
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: PAD; Critical Limb Ischemia; Atherosclerotic Ischemic Disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PB-MNC therapy (Active Comparator): The patientsin PB-MNC therapy group will be injected with G-CSF mobilized PB-MNC into calf or thigh muscle of ischemic limb and Aspirin 81 mg/day and supportive treatment including wound care and pain killer drug.
  Interventions: Procedure: PB-MNC therapy
- No PB-MNC therapy (Active Comparator): In patients in No PB-MNC therapy, they will receive aspirin 81 mg/day and supportive treatment including wound care and pain killer drug.
  Interventions: Drug: No-PB-MNC therapy

INTERVENTIONS:
Procedure: PB-MNC therapy — The patients will receive subcutaneous injection of Granulocyte colony stimulating factor (G-CSF) for 3 day. The mononuclear cell will be collected by blood cell separator. The 120 cc of cell solution will be injected into calf or thigh of ischemic limb (1cc per site) with needle no. 25 gauge. Patients will receive ASA 81 mg once daily and wound care and pain killer drug
  Arms: PB-MNC therapy
Drug: No-PB-MNC therapy — Patients will receive ASA 81 mg once daily and wound care and pain killer drug
  Arms: No PB-MNC therapy

SUMMARY:
This study will investigate the efficacy of G-CSF mobilized mononuclear cell injection of patients with PAD who presented with no-option CLI. Forty no-option CLI patients who presented with rest pain, non-healing ischemic ulcer or gangrene will be randomized into 2 groups. The control group will be treated by medication and supportive treatment. The experiment group will be injected G-CSF mobilized mononuclear cell ,medication. Amputation free survival,Ankle brachial index(ABI), Toe brachial index (TBI) and transcutaneous oxygen measurement will be evaluated at the day of randomization, 1 , 3, 6 and 12 months.

DETAILED DESCRIPTION:
This study will investigate the efficacy of G-CSF mobilized mononuclear cell injection of patients with PAD who presented with no-option CLI. Forty no-option CLI patients who presented with rest pain, non-healing ischemic ulcer or gangrene will be randomized into 2 groups. The control group will be treated by medication and supportive treatment. The experiment group will be injected G-CSF mobilized mononuclear cell ,medication. Ankle brachial index(ABI), Toe brachial index (TBI) and transcutaneous oxygen measurement will be evaluated at the day of randomization, 1 , 3, 6 and 12 months in the control group and day of randomization, 1 , 3, 6 and 12 months after injection of PB-MNC in the experiment group. Amputation free survival will be evaluated at , 1 , 3, 6 and 12 months after PB-MNC therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with no-option CLI who presented with rest pain , non-healing ischemic ulcer and toe gangrene for 3 months

Exclusion Criteria:

* Recent myocardial infarction
* Severe valvular heart disease
* After organ transplantation
* Cardiomyopthy( EF< 25%)
* Liver failure
* Coagulopathy
* HIV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Amputation free survival | 3 month
  Rate of non amputated limb

SECONDARY OUTCOMES:
Amputation free survival | 1,6,12 month
  Rate of non amputated limb
Ankle brachial index (ABI) | 1,3,6,12 month
  Ankle brachial indexThe Ankle Brachial Index (ABI) is the systolic pressure at the ankle, divided by the systolic pressure at the arm. It has been shown to be a specific and sensitive metric for the diagnosis of Peripheral Arterial Disease (PAD)
Toe brachial index (TBI) | 1,3,6,12 month
  Toe brachial indexThe toe brachial index is the ratio between toe pressure and the highest of the two brachial pressures
Transcutaneous oxygen measurement (TCOM) | 1,3,6,12 month
  Transcutaneous oxygen measurement
36-Item Short Form Health Survey (SF36) | 1,3,6,12 month
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Nuttawut SERMSATHANASAWADI, Principal Investigator — Mahidol University
Locations (1):
- Vascular Surgery, Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No